CLINICAL TRIAL: NCT04102306
Title: Assessing Motor Imagery Using the Tongue and Mouth Imagery Questionnaire (TMIQ) in Patients With Temporomandibular Disorder and Healthy Control Subjects: a Reliability and Construct Validity Study
Brief Title: Assessing Motor Imagery Ability of Tongue and Mouth in Subjects With and With no Temporomandibular Disorders
Acronym: TMIQ
Status: Completed | Type: Observational
Sponsor: Cabinet de Kinesitherapie SCM Saint-Alexandre (Industry)
Collaborators: University of Lyon (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: TMIQ
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-09

CONDITIONS: Temporomandibular Disorder; Motor Imagery
Keywords: orofacial myotherapies;; physical therapy;; assessment;; questionnaire validation
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular disorder group (TMD): Patients with temporomandibular disorder coming at the Cabinet Saint Alexandre for orofacial rehabilitation.
  Test 1: passation of the KVIQ questionnaire, followed by the passation of the TMIQ during a rehabilitation session supervised by the physical therapist (PT) Test 2: passation of the TMIQ during the next rehabilitation session supervised by the same PT(interval between PT session 1 and 2 is a maximum of 45 days).
  Questionnaires were performed during the course of the patient rehabilitation that was instructed not to perform imagined movement during the interval.
  Interventions: Other: reliability and validity construct of the TMIQ
- Control healthy group (CTL): Healthy individuals with no temporomandibular disorder (i.e., no orofacial medical consultation or rehabilitation) aged-matched and gender-matched to TMD group.
  Test 1: passation of the KVIQ questionnaire, followed by the passation of the TMIQ during a session supervised by the physical therapist (PT) Test 2: passation of the TMIQ during the next session supervised by the same PT(interval between PT session 1 and 2 is a maximum of 8 days).
  Questionnaires were performed with no additional rehabilitation and participants were instructed not to perform imagined movement during the interval.
  Interventions: Other: reliability and validity construct of the TMIQ

INTERVENTIONS:
Other: reliability and validity construct of the TMIQ — comparison of the TMIQ to the gold-standard questionnaire (KVIQ) and test-retest

SUMMARY:
Temporomandibular disorder (TMD) is the symptomatic expression of a muscular or an articular impairment at the manducatory tract. TMD affects between 30 to 65% of the population with a higher prevalence for young women. The patients with DTM report a decrease of their personal, social and professional quality of life. Treatment usually relies on physical therapy. Among the different technics that can be used in physical therapy, there is growing evidence advocating the efficacy of using motor imagery (i.e. imagining a movement with no concomitant physical execution) during rehabilitation. It has also been shown that the benefits of practicing motor imagery depend on the ability (i.e., the higher the ability, the greater the benefits). However, there is no investigation of the motor imagery ability of the tongue and mouth movements conditioning the use of motor imagery during TMD rehabilitation. The objective of the study is to investigate the ability of imagining tongue and mouth movements using the Tongue and Mouth Imagery Questionnaire (TMIQ) as compare to the gold-standard Kinesthetic and Visual Imagery Questionnaire (KVIQ - Malouin et al., 2007).

DETAILED DESCRIPTION:
Principal objective:

Assess the validity construct of the Tongue and Mouth Imagery Questionnaire (TMIQ) as compare to the gold-standard Kinesthetic and Visual Imagery Questionnaire (KVIQ - Malouin et al., 2007), both measuring the motor imagery vividness.

Secondary objectives:

1. Assess the reliability of the TMIQ using a test-retest.
2. Assess the temporal coupling (i.e., the ratio between imagined and physically practiced movement) and compare these ratios for the TMIQ and KVIQ.
3. Investigate the effect of TMD by comparing the vividness scores of TMIQ for respectively subject with and with no TMD.
4. Investigate the effect of TMD by comparing the vividness scores of KVIQ for respectively subject with and with no TMD.
5. Investigate the effect of TMD by comparing the temporal coupling scores of TMIQ for respectively subject with and with no TMD.
6. Investigate the effect of TMD by comparing the temporal coupling scores of KVIQ for respectively subject with and with no TMD.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* A voluntary individual who has given informed consent after receiving clear, fair and appropriate information about the study.

For DTM group participants

* inclusion during the DTM rehabilitation in the physical therapy firm "Cabinet Saint Alexandre".
* beneficiary of the social security scheme

Exclusion Criteria:

* The presence of a short tongue brake (Marchesan, 2005)
* Lingual immaturity evaluated by the Tardieu test (Jouannaud et al. 1972)
* Patients who had orthognathic surgery within 6 months post- operative, or facial fractures according to the same deadlines
* The presence of peripheral facial palsy
* Current participation in another research whose objective would be the evaluation of a therapeutic, drug or not, introducing an experimental bias.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 47 participants with DTM 47 participants with no DTM (healthy control) age-matched and gender-matched to participants with DTM.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
vividness score of imagined movements of the TMIQ for the DTM group | at study inclusion, i.e day 1
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the TMIQ for the DTM group
vividness score of imagined movements of the TMIQ for the CTL group | at study inclusion, i.e day 1
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the TMIQ for the DTM group
vividness score of imagined movements of the KVIQ for the DTM group | at study inclusion, i.e day 1
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the KVIQ for the DTM group
vividness score of imagined movements of the KVIQ for the CTL group | at study inclusion, i.e day 1
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the KVIQ for the DTM group

SECONDARY OUTCOMES:
vividness score of imagined movements of the TMIQ for the DTM group | at study completion, between 8 days to 45 days after inclusion
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the TMIQ for the DTM group
vividness score of imagined movements of the TMIQ for the CTL group | at study completion, between 8 days to 45 days after inclusion
  Averaged vividness score (using a 5-point likert scale, 1=minimum vividness, 5=maximal vividness) for the TMIQ for the DTM group
Temporal coupling to imagined movements of the TMIQ for the DTM group | at study completion, between 8 days to 45 days after inclusion
  Computation of ratio between imagined and physically practiced movements measured during the TMIQ for the DTM group
Temporal coupling to imagined movements of the TMIQ for the CTL group | at study inclusion, i.e day 1
  Computation of ratio between imagined and physically practiced movements measured during the TMIQ for the DTM group
Temporal coupling to imagined movements of the TMIQ for the CTL group | at study completion, between 8 days to 45 days after inclusion
  Computation of ratio between imagined and physically practiced movements measured during the TMIQ for the DTM group

OTHER OUTCOMES:
mental representation of the maximal opening of the mouth for the DTM group | at study inclusion, i.e day 1
  comparison of the score (5-point likert Scale, 1= minimal opening, 5=maximal opening) self-reported by the participant after imagination of maximal mouth opening as compared to the score of the physical therapist after the physical execution of mouth opening by the participant during the TMIQ for the DTM group
mental representation of the maximal opening of the mouth for the CTL group | at study inclusion, i.e day 1
  comparison of the score (5-point likert Scale, 1= minimal opening, 5=maximal opening) self-reported by the participant after imagination of maximal mouth opening as compared to the score of the physical therapist after the physical execution of mouth opening by the participant during the TMIQ for the CTL group
Accuracy of tongue pointing against the wood examination stick for the DTM group | at study inclusion, i.e day 1
  Measure the surface of the tongue print after that participant was requested to point as accurately as possible while keeping the tongue sharp against the wood examination stick for the DTM group
Accuracy of tongue pointing against the wood examination stick for the CTL group | at study inclusion, i.e day 1
  Measure the surface of the tongue print after that participant was requested to point as accurately as possible while keeping the tongue sharp against the wood examination stick for the CTL group

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Alvarado-Faysse, PT, Principal Investigator — Cabinet de kinésithérapie Saint Alexandre
Locations (1):
- Cabinet Saint Alexandre, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alvarado C, Arminjon A, Damieux-Verdeaux C, Lhotte C, Condemine C, Cousin AS, Sigaux N, Bouletreau P, Mateo S. Impaired tongue motor control after temporomandibular disorder: A proof-of-concept case-control study of tongue print. Clin Exp Dent Res. 2022 Apr;8(2):529-536. doi: 10.1002/cre2.549. Epub 2022 Feb 27. PMID 35220688